CLINICAL TRIAL: NCT03923933
Title: Chlortalidone and Bumetanide in Advanced Chronic Kidney Disease: HEBE-CKD Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital General de México Dr. Eduardo Liceaga (Other Government)
Responsible Party: Principal Investigator, Fabio Solis-Jimenez, Principal Investigator, Hospital General de México Dr. Eduardo Liceaga
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DI/19/105-B/03/018
Record Dates: First submitted 2019-04-18; First posted 2019-04-23 (Actual); Results first posted 2020-03-10 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Renal Insufficiency, Chronic
Keywords: Diuretics; Bumetanide; Chlorthalidone; Chronic Kidney Disease; Volume Overload
MeSH Terms: conditions — Renal Insufficiency, Chronic; Edema | interventions — Chlorthalidone; Bumetanide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): This group will receive 3 milligrams of bumetanide per day for a week plus placebo (starch) that will simulate the chlorthalidone dose of the treatment group. In case the dose is well tolerated, the dose of bumetanide will be increased to 4 milligrams per day.
  Interventions: Drug: Bumetanide
- Treatment grup (Experimental): This group will receive 3 milligrams of bumetanide plus 50 milligrams of chlorthalidone per day, for a week. If the dose is well tolerated, it will be increased to 4 milligrams of bumetanide and 100 milligrams of chlorthalidone per day.
  Interventions: Drug: Chlorthalidone; Drug: Bumetanide

INTERVENTIONS:
Drug: Chlorthalidone — Chlorthalidone
  Arms: Treatment grup
Drug: Bumetanide — Bumetanide

SUMMARY:
This study aims to demonstrate the possible benefit of a treatment based on double diuretic in patients with chronic kidney disease and severely impaired glomerular filtration rate. This is based on previous observations where the investigators found that volume overload is a frequent condition within this population and is strongly linked to an increase in morbidity and mortality. The investigators consider that this therapy could be beneficial given that most of these patients are treated with loop diuretics, however, with the passage of time, adaptive changes in the distal nephron occur that promote a decrease in the treatment effect. In this sense, thiazide diuretics at appropriate doses could 'break' the resistance, since their mechanism of action antagonizes the resistance mechanism. Unfortunately, to this day, this treatment has not been fully evaluated. Particularly in this type of population.

The investigators developed a study proposed as a double blind randomized clinical trial, where the population will be divided into two groups. A group will be given the standard treatment based on loop diuretic (bumetanide), while the other group will receive the intervention (bumetanide plus chlorthalidone). After a 30-day follow-up period, the results will be measured.

With respect to the effectiveness of the treatment, the decrease in volume overload by bioimpedance will be measured. While the occurrence of adverse effects during the same monitoring period will be observed.

ELIGIBILITY:
Inclusion Criteria:

* glomerular filtration rate less than 30 ml / min / 1.73m
* Without replacement therapy (dialysis or hemodialysis)
* Volume overload
* At least 100 ml per day of residual diuresis
* Use of a loop diuretic for at least one month

Exclusion Criteria:

* Allergies known to diuretics
* Patients with severe infections
* Patients with hemodynamic instability
* Amputees
* Patients with cognitive impairment
* Patients with acute renal failure
* Patients with graft loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2019-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Solis-Jimenez, M.D., Principal Investigator — Hospital General de México Dr. Eduardo Liceaga
Locations (1):
- Hospital General de Mexico, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bello AK, Levin A, Tonelli M, Okpechi IG, Feehally J, Harris D, Jindal K, Salako BL, Rateb A, Osman MA, Qarni B, Saad S, Lunney M, Wiebe N, Ye F, Johnson DW. Assessment of Global Kidney Health Care Status. JAMA. 2017 May 9;317(18):1864-1881. doi: 10.1001/jama.2017.4046. PMID 28430830
- [Background] Neuen BL, Chadban SJ, Demaio AR, Johnson DW, Perkovic V. Chronic kidney disease and the global NCDs agenda. BMJ Glob Health. 2017 Jul 6;2(2):e000380. doi: 10.1136/bmjgh-2017-000380. eCollection 2017. No abstract available. PMID 29225940
- [Background] Levey AS, Coresh J. Chronic kidney disease. Lancet. 2012 Jan 14;379(9811):165-80. doi: 10.1016/S0140-6736(11)60178-5. Epub 2011 Aug 15. PMID 21840587
- [Background] van de Luijtgaarden MW, Noordzij M, van Biesen W, Couchoud C, Cancarini G, Bos WJ, Dekker FW, Gorriz JL, Iatrou C, Wanner C, Finne P, Stojceva-Taneva O, Cala S, Stel VS, Tomson C, Jager KJ. Conservative care in Europe--nephrologists' experience with the decision not to start renal replacement therapy. Nephrol Dial Transplant. 2013 Oct;28(10):2604-12. doi: 10.1093/ndt/gft287. Epub 2013 Sep 7. PMID 24013682
- [Background] Morton RL, Turner RM, Howard K, Snelling P, Webster AC. Patients who plan for conservative care rather than dialysis: a national observational study in Australia. Am J Kidney Dis. 2012 Mar;59(3):419-27. doi: 10.1053/j.ajkd.2011.08.024. Epub 2011 Oct 20. PMID 22014401
- [Background] Wong SPY, Hebert PL, Laundry RJ, Hammond KW, Liu CF, Burrows NR, O'Hare AM. Decisions about Renal Replacement Therapy in Patients with Advanced Kidney Disease in the US Department of Veterans Affairs, 2000-2011. Clin J Am Soc Nephrol. 2016 Oct 7;11(10):1825-1833. doi: 10.2215/CJN.03760416. Epub 2016 Sep 22. PMID 27660306
- [Background] Davison SN, Levin A, Moss AH, Jha V, Brown EA, Brennan F, Murtagh FE, Naicker S, Germain MJ, O'Donoghue DJ, Morton RL, Obrador GT; Kidney Disease: Improving Global Outcomes. Executive summary of the KDIGO Controversies Conference on Supportive Care in Chronic Kidney Disease: developing a roadmap to improving quality care. Kidney Int. 2015 Sep;88(3):447-59. doi: 10.1038/ki.2015.110. Epub 2015 Apr 29. PMID 25923985
- [Background] Verberne WR, Dijkers J, Kelder JC, Geers ABM, Jellema WT, Vincent HH, van Delden JJM, Bos WJW. Value-based evaluation of dialysis versus conservative care in older patients with advanced chronic kidney disease: a cohort study. BMC Nephrol. 2018 Aug 16;19(1):205. doi: 10.1186/s12882-018-1004-4. PMID 30115028
- [Background] Murtagh FE, Addington-Hall JM, Edmonds PM, Donohoe P, Carey I, Jenkins K, Higginson IJ. Symptoms in advanced renal disease: a cross-sectional survey of symptom prevalence in stage 5 chronic kidney disease managed without dialysis. J Palliat Med. 2007 Dec;10(6):1266-76. doi: 10.1089/jpm.2007.0017. PMID 18095805
- [Background] Thomas R, Kanso A, Sedor JR. Chronic kidney disease and its complications. Prim Care. 2008 Jun;35(2):329-44, vii. doi: 10.1016/j.pop.2008.01.008. PMID 18486718
- [Background] Hung SC, Lai YS, Kuo KL, Tarng DC. Volume overload and adverse outcomes in chronic kidney disease: clinical observational and animal studies. J Am Heart Assoc. 2015 May 5;4(5):e001918. doi: 10.1161/JAHA.115.001918. PMID 25944876
- [Background] Titze J. Interstitial fluid homeostasis and pressure: news from the black box. Kidney Int. 2013 Nov;84(5):869-71. doi: 10.1038/ki.2013.287. PMID 24172732
- [Background] Yatime L, Laursen M, Morth JP, Esmann M, Nissen P, Fedosova NU. Structural insights into the high affinity binding of cardiotonic steroids to the Na+,K+-ATPase. J Struct Biol. 2011 May;174(2):296-306. doi: 10.1016/j.jsb.2010.12.004. Epub 2010 Dec 21. PMID 21182963
- [Background] Khalaf FK, Dube P, Mohamed A, Tian J, Malhotra D, Haller ST, Kennedy DJ. Cardiotonic Steroids and the Sodium Trade Balance: New Insights into Trade-Off Mechanisms Mediated by the Na(+)/K(+)-ATPase. Int J Mol Sci. 2018 Aug 30;19(9):2576. doi: 10.3390/ijms19092576. PMID 30200235
- [Background] Akchurin OM, Kaskel F. Update on inflammation in chronic kidney disease. Blood Purif. 2015;39(1-3):84-92. doi: 10.1159/000368940. Epub 2015 Jan 20. PMID 25662331
- [Background] Maruta Y, Hasegawa T, Yamakoshi E, Nishiwaki H, Koiwa F, Imai E, Hishida A. Association between serum Na-Cl level and renal function decline in chronic kidney disease: results from the chronic kidney disease Japan cohort (CKD-JAC) study. Clin Exp Nephrol. 2019 Feb;23(2):215-222. doi: 10.1007/s10157-018-1631-x. Epub 2018 Aug 24. PMID 30168046
- [Background] Khan YH, Sarriff A, Adnan AS, Khan AH, Mallhi TH. Chronic Kidney Disease, Fluid Overload and Diuretics: A Complicated Triangle. PLoS One. 2016 Jul 21;11(7):e0159335. doi: 10.1371/journal.pone.0159335. eCollection 2016. PMID 27442587
- [Background] Arikan AA, Zappitelli M, Goldstein SL, Naipaul A, Jefferson LS, Loftis LL. Fluid overload is associated with impaired oxygenation and morbidity in critically ill children. Pediatr Crit Care Med. 2012 May;13(3):253-8. doi: 10.1097/PCC.0b013e31822882a3. PMID 21760565
- [Background] Hassinger AB, Wald EL, Goodman DM. Early postoperative fluid overload precedes acute kidney injury and is associated with higher morbidity in pediatric cardiac surgery patients. Pediatr Crit Care Med. 2014 Feb;15(2):131-8. doi: 10.1097/PCC.0000000000000043. PMID 24366508
- [Background] Magee G, Zbrozek A. Fluid overload is associated with increases in length of stay and hospital costs: pooled analysis of data from more than 600 US hospitals. Clinicoecon Outcomes Res. 2013 Jun 26;5:289-96. doi: 10.2147/CEOR.S45873. Print 2013. PMID 23836999
- [Background] Vaara ST, Korhonen AM, Kaukonen KM, Nisula S, Inkinen O, Hoppu S, Laurila JJ, Mildh L, Reinikainen M, Lund V, Parviainen I, Pettila V; FINNAKI Study Group. Fluid overload is associated with an increased risk for 90-day mortality in critically ill patients with renal replacement therapy: data from the prospective FINNAKI study. Crit Care. 2012 Oct 17;16(5):R197. doi: 10.1186/cc11682. PMID 23075459
- [Background] Di Lullo L, Gorini A, Russo D, Santoboni A, Ronco C. Left Ventricular Hypertrophy in Chronic Kidney Disease Patients: From Pathophysiology to Treatment. Cardiorenal Med. 2015 Oct;5(4):254-66. doi: 10.1159/000435838. Epub 2015 Jul 15. PMID 26648942
- [Background] Ekinci C, Karabork M, Siriopol D, Dincer N, Covic A, Kanbay M. Effects of Volume Overload and Current Techniques for the Assessment of Fluid Status in Patients with Renal Disease. Blood Purif. 2018;46(1):34-47. doi: 10.1159/000487702. Epub 2018 Apr 12. PMID 29649794
- [Background] Collins AJ, Foley RN, Gilbertson DT, Chen SC. United States Renal Data System public health surveillance of chronic kidney disease and end-stage renal disease. Kidney Int Suppl (2011). 2015 Jun;5(1):2-7. doi: 10.1038/kisup.2015.2. PMID 26097778
- [Background] Chang ST, Chen CL, Chen CC, Lin FC, Wu D. Enhancement of quality of life with adjustment of dry weight by echocardiographic measurement of inferior vena cava diameter in patients undergoing chronic hemodialysis. Nephron Clin Pract. 2004;97(3):c90-7. doi: 10.1159/000078636. PMID 15292685
- [Background] Andreucci M, Russo D, Fuiano G, Minutolo R, Andreucci VE. Diuretics in renal failure. Miner Electrolyte Metab. 1999 Jan-Apr;25(1-2):32-8. doi: 10.1159/000057416. PMID 10207256
- [Background] Wilcox CS. New insights into diuretic use in patients with chronic renal disease. J Am Soc Nephrol. 2002 Mar;13(3):798-805. doi: 10.1681/ASN.V133798. PMID 11856788
- [Background] National Kidney Foundation. K/DOQI clinical practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Am J Kidney Dis. 2002 Feb;39(2 Suppl 1):S1-266. No abstract available. PMID 11904577
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; National Heart, Lung, and Blood Institute Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure; National High Blood Pressure Education Program Coordinating Committee. The Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure: the JNC 7 report. JAMA. 2003 May 21;289(19):2560-72. doi: 10.1001/jama.289.19.2560. Epub 2003 May 14. PMID 12748199
- [Background] Roberts MA. Commentary on the KDIGO Clinical Practice Guideline for the management of blood pressure in chronic kidney disease. Nephrology (Carlton). 2014 Jan;19(1):53-5. doi: 10.1111/nep.12168. No abstract available. PMID 24341660
- [Background] James PA, Oparil S, Carter BL, Cushman WC, Dennison-Himmelfarb C, Handler J, Lackland DT, LeFevre ML, MacKenzie TD, Ogedegbe O, Smith SC Jr, Svetkey LP, Taler SJ, Townsend RR, Wright JT Jr, Narva AS, Ortiz E. 2014 evidence-based guideline for the management of high blood pressure in adults: report from the panel members appointed to the Eighth Joint National Committee (JNC 8). JAMA. 2014 Feb 5;311(5):507-20. doi: 10.1001/jama.2013.284427. PMID 24352797
- [Background] Hoorn EJ, Ellison DH. Diuretic Resistance. Am J Kidney Dis. 2017 Jan;69(1):136-142. doi: 10.1053/j.ajkd.2016.08.027. Epub 2016 Nov 1. PMID 27814935
- [Background] Bowman BN, Nawarskas JJ, Anderson JR. Treating Diuretic Resistance: An Overview. Cardiol Rev. 2016 Sep-Oct;24(5):256-60. doi: 10.1097/CRD.0000000000000116. PMID 27465540
- [Background] Ellison DH, Felker GM. Diuretic Treatment in Heart Failure. N Engl J Med. 2017 Nov 16;377(20):1964-1975. doi: 10.1056/NEJMra1703100. No abstract available. PMID 29141174
- [Background] Knepper MA. Systems biology of diuretic resistance. J Clin Invest. 2015 May;125(5):1793-5. doi: 10.1172/JCI81505. Epub 2015 Apr 20. PMID 25893597
- [Background] Shahin MH, Johnson JA. Mechanisms and pharmacogenetic signals underlying thiazide diuretics blood pressure response. Curr Opin Pharmacol. 2016 Apr;27:31-7. doi: 10.1016/j.coph.2016.01.005. Epub 2016 Feb 10. PMID 26874237
- [Background] Yugar LBT, Moreno B, Moreno H, Vilela-Martin JF, Yugar-Toledo JC. Do thiazide diuretics reduce central systolic blood pressure in hypertension? J Clin Hypertens (Greenwich). 2018 Jan;20(1):133-135. doi: 10.1111/jch.13134. Epub 2017 Nov 6. No abstract available. PMID 29106774
- [Background] REUBI FC, COTTIER PT. Effects of reduced glomerular filtration rate on responsiveness to chlorothiazide and mercurial diuretics. Circulation. 1961 Feb;23:200-10. doi: 10.1161/01.cir.23.2.200. No abstract available. PMID 13740990
- [Background] Bennett WM, Porter GA. Efficacy and safety of metolazone in renal failure and the nephrotic syndrome. J Clin Pharmacol. 1973 Aug-Sep;13(8):357-64. doi: 10.1002/j.1552-4604.1973.tb00224.x. No abstract available. PMID 4579972
- [Background] Dargie HJ, Allison ME, Kennedy AC, Gray MJ. High dosage metolazone in chronic renal failure. Br Med J. 1972 Oct 28;4(5834):196-8. doi: 10.1136/bmj.4.5834.196. PMID 5082545
- [Background] Craswell PW, Ezzat E, Kopstein J, Varghese Z, Moorhead JF. Use of metolazone, a new diuretic, in patients with renal disease. Nephron. 1974;12(1):63-73. doi: 10.1159/000180257. No abstract available. PMID 4838012
- [Background] Dargie HJ, Allison ME, Kennedy AC, Gray MJ. Efficacy of metolazone in patients with renal edema. Clin Nephrol. 1974;2(4):157-60. No abstract available. PMID 4847130
- [Background] Wollam GL, Tarazi RC, Bravo EL, Dustan HP. Diuretic potency of combined hydrochlorothiazide and furosemide therapy in patients with azotemia. Am J Med. 1982 Jun;72(6):929-38. doi: 10.1016/0002-9343(82)90854-3. PMID 7046434
- [Background] Fliser D, Schroter M, Neubeck M, Ritz E. Coadministration of thiazides increases the efficacy of loop diuretics even in patients with advanced renal failure. Kidney Int. 1994 Aug;46(2):482-8. doi: 10.1038/ki.1994.298. PMID 7967362
- [Background] Knauf H, Mutschler E. Diuretic effectiveness of hydrochlorothiazide and furosemide alone and in combination in chronic renal failure. J Cardiovasc Pharmacol. 1995 Sep;26(3):394-400. doi: 10.1097/00005344-199509000-00008. PMID 8583780
- [Background] Dussol B, Moussi-Frances J, Morange S, Somma-Delpero C, Mundler O, Berland Y. A randomized trial of furosemide vs hydrochlorothiazide in patients with chronic renal failure and hypertension. Nephrol Dial Transplant. 2005 Feb;20(2):349-53. doi: 10.1093/ndt/gfh650. Epub 2004 Dec 22. PMID 15615808
- [Background] Dussol B, Moussi-Frances J, Morange S, Somma-Delpero C, Mundler O, Berland Y. A pilot study comparing furosemide and hydrochlorothiazide in patients with hypertension and stage 4 or 5 chronic kidney disease. J Clin Hypertens (Greenwich). 2012 Jan;14(1):32-7. doi: 10.1111/j.1751-7176.2011.00564.x. Epub 2011 Dec 9. PMID 22235821
- [Background] Agarwal R, Sinha AD, Pappas MK, Ammous F. Chlorthalidone for poorly controlled hypertension in chronic kidney disease: an interventional pilot study. Am J Nephrol. 2014;39(2):171-82. doi: 10.1159/000358603. Epub 2014 Feb 11. PMID 24526255
- [Background] Cirillo M, Marcarelli F, Mele AA, Romano M, Lombardi C, Bilancio G. Parallel-group 8-week study on chlorthalidone effects in hypertensives with low kidney function. Hypertension. 2014 Apr;63(4):692-7. doi: 10.1161/HYPERTENSIONAHA.113.02793. Epub 2014 Jan 6. PMID 24396024
- [Derived] Solis-Jimenez F, Perez-Navarro LM, Cabrera-Barron R, Chida-Romero JA, Martin-Alemany G, Dehesa-Lopez E, Madero M, Valdez-Ortiz R. Effect of the combination of bumetanide plus chlorthalidone on hypertension and volume overload in patients with chronic kidney disease stage 4-5 KDIGO without renal replacement therapy: a double-blind randomized HEBE-CKD trial. BMC Nephrol. 2022 Sep 20;23(1):316. doi: 10.1186/s12882-022-02930-4. PMID 36127661

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the nephrology clinic in the Hospital General de México, between May and August 2019. All those with stage 4-5 chronic kidney disease, who had chronic use of loop diuretics and hypertension, were invited to perform an impedance measurement. Those with volume overload were invited to participate in the protocol.
Period: Overall Study
Arm/Group | Placebo | Treatment Grup
Started | 17 | 17
Completed | 16 | 16
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Treatment Grup | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (8.1) | 54.8 (10) | 57.2 (9.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 4 | 6 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Mexico | 16 | 16 | 32
Total body water [Median (Full Range); unit: liters] | 33.1 [20 to 53.7] | 32.7 [23.4 to 70.6] | 33.1 [20 to 70.6]
Extracellular water [Median (Full Range); unit: liters] | 16.2 [10.7 to 25.8] | 16.4 [12.8 to 35.7] | 16.3 [10.7 to 35.7]
Extracellular water/Total Body Water [Mean (Standard Deviation); unit: percentage] | 50.9 (3.5) | 50 (3.6) | 50.4 (3.5)
systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 146.8 (18.2) | 142 (22.6) | 144.6 (20.3)
diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 77.8 (11.3) | 81.8 (10.9) | 79.7 (11.1)
Mean arterial pressure [Mean (Standard Deviation); unit: mmHg] | 100.6 (12.8) | 102.1 (10.9) | 101 (12.7)
serum creatinine [Median (Full Range); unit: mg/dL] | 3.5 [1.9 to 15] | 3.6 [1.8 to 16.6] | 3.6 [1.8 to 16.6]
serum urea [Median (Full Range); unit: mg/dL] | 124 [85.4 to 269] | 125 [57.9 to 244.9] | 125 [57.9 to 269]
glomerular filtration rate [Mean (Standard Deviation); unit: ml/min/1.73m2] | 15.69 (7.64) | 16.52 (8.76) | 16.1 (8.14)
Cause of chronic kidney disease [Count of Participants; unit: Participants]
  Diabetes | 11 | 11 | 22
  Hypertension | 1 | 1 | 2
  Lupus | 1 | 0 | 1
  Unknown | 3 | 4 | 7
Seric sodium [Mean (Standard Deviation); unit: meq/l] | 138.3 (4.3) | 137.4 (4.9) | 137.9 (4.6)
serum potassium [Mean (Standard Deviation); unit: meq/l] | 5.1 (0.74) | 5.3 (0.64) | 5.2 (0.68)
Urinary sodium [Mean (Standard Deviation); unit: meq/l] | 64.7 (23.4) | 62.7 (20.6) | 63.7 (21.6)
Urinary chlorine [Mean (Standard Deviation); unit: meq/l] | 60.2 (27.4) | 62.3 (18.6) | 61.2 (23.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Body Water
Description: Measured by bioelectrical impedance analysis, compared to the initial measurement
Time Frame: Change from Basal to day 28
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Treatment Grup
Number analyzed (Participants) | 16 | 16
litres | -0.075 (1.78) | -4.36 (3.29)
Statistical Analysis 1: Comparison: Placebo vs Treatment Grup; Test type: Superiority; p < 0.001, ANOVA; anova repeated measures

2. Secondary Outcome: Change in Mean Arterial Pressure
Description: decrease in blood pressure compared wit baseline measure (mmhg)
Time Frame: Change from Basal to day 28
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Treatment Grup
Number analyzed (Participants) | 16 | 16
mmHg | -5.4 (14.3) | -18.1 (8.7)
Statistical Analysis 1: Comparison: Placebo vs Treatment Grup; Test type: Superiority; p = 0.006, ANOVA; Repeated Measures

3. Secondary Outcome: Change in the Fractional Excretion of Sodium
Description: Increase in the fractional excretion of sodium compared with the baseline measure
Time Frame: Change from Basal to day 28
Measure: Mean (Standard Deviation); unit: percentage of sodium excreted
Arm/Group | Placebo | Treatment Grup
Number analyzed (Participants) | 16 | 16
percentage of sodium excreted | -0.348 (3.48) | 0.598 (2.29)
Statistical Analysis 1: Comparison: Placebo vs Treatment Grup; Test type: Superiority; p = 0.371, ANOVA

4. Secondary Outcome: Change in Extracellular Water
Description: Decrease in extracellular water measured by bioelectrical impedance analysis
Time Frame: Change from Basal to day 28
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Treatment Grup
Number analyzed (Participants) | 16 | 16
litres | -0.15 (1.2) | 2.55 (1.1)
Statistical Analysis 1: Comparison: Placebo vs Treatment Grup; Test type: Superiority; p < 0.001, ANOVA

5. Secondary Outcome: Change in Extracellular Water / Total Body Water Ratio
Description: Decrease in extracellular water / total body water ratio measured by bioelectrical impedance analysis
Time Frame: Change from Basal to day 28
Measure: Mean (Standard Deviation); unit: percentage of ECW/TBW
Arm/Group | Placebo | Treatment Grup
Number analyzed (Participants) | 16 | 16
percentage of ECW/TBW | -0.24 (1.42) | -2.92 (4.76)

6. Secondary Outcome: Change in Systolic Blood Pressure
Time Frame: Change from Basal to day 28
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Treatment Grup
Number analyzed (Participants) | 16 | 16
mmHg | -10 (23.3) | -26.1 (15.3)
Statistical Analysis 1: Comparison: Placebo vs Treatment Grup; Test type: Superiority; p = 0.028, ANOVA

7. Secondary Outcome: Change in Diastolic Blood Pressure
Time Frame: Change from Basal to day 28
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Treatment Grup
Number analyzed (Participants) | 16 | 16
mmHg | -3.4 (11.9) | -13.5 (10.7)
Statistical Analysis 1: Comparison: Placebo vs Treatment Grup; Test type: Superiority; p = 0.018, ANOVA

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Placebo | Treatment Grup
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 1/16
Other Adverse Events (participants affected / at risk) | 4/16 | 11/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=16) | Treatment Grup (N=16)
Major adverse cardiovascular events (Cardiac disorders) | 0 (0) | 1 (1) — Nonfatal stroke, nonfatal myocardial infarction, and cardiovascular death
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=16) | Treatment Grup (N=16)
Creatinine Increase (Renal and urinary disorders) | 4 (4) | 11 (11) — increase in serum creatinine levels greater than 0.3 mg / dl compared to baseline
Hyponatremia (Renal and urinary disorders) | 1 (1) | 2 (2) — Seric sodium less than 129 meq / liter
hypokalemia (Renal and urinary disorders) | 0 (0) | 2 (2) — Seric potassium less than 3.5 meq/litre
hyperuricemia (Renal and urinary disorders) | 4 (4) | 4 (4) — Seric uric acid greater than 8 mg/dl

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/33/NCT03923933/Prot_SAP_000.pdf